CLINICAL TRIAL: NCT03923231
Title: Investigation of the Pharmacokinetics of Atazanavir in Pregnant Women, Individuals at Extremes of BMI, Children, and Adolescents: An Observational Study Nested Within the VirTUAL Consortium
Brief Title: Pharmacokinetics of Atazanavir in Special Populations
Acronym: VirTUAL WP5
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Makerere University (Other); Joint Clinical Research Centre- Kampala (Unknown); Desmond Tutu HIV Foundation (Other); University of Cape Town (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) - funder (Unknown)
Responsible Party: Principal Investigator, Catriona Waitt, Senior Lecturer in Clinical Pharmacology, University of Liverpool
Other Study IDs: VirTUAL WP5
Record Dates: First submitted 2019-04-15; First posted 2019-04-22 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: HIV/AIDS; Tuberculosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis | interventions — Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Children <5 years: Children under the age of 5 years who are receiving atazanavir as part of clinical care
  Interventions: Drug: Atazanavir 250 mg / ritonavir 80 mg
- Children 6-11: Children aged 6-11 years who are receiving atazanavir as part of clinical care
  Interventions: Drug: Atazanavir 250 mg / ritonavir 80 mg
- Adolescents 12-17: Adolescents aged 12-17 years who are receiving atazanavir as part of clinical care
  Interventions: Drug: Atazanavir 300mg/ Ritonavir 100 mg once daily
- Pregnant women: Women who are at least 20 weeks gestation, who are receiving atazanavir as part of clinical care
  Interventions: Drug: Atazanavir 300mg/ Ritonavir 100 mg once daily
- BMI < 18.5: Adults with a BMI of <18.5 kg/m2 who are receiving atazanavir as part of clinical care
  Interventions: Drug: Atazanavir 300mg/ Ritonavir 100 mg once daily
- BMI >30: Adults with a BMI of >30 kg/m2 who are receiving atazanavir as part of clinical care
  Interventions: Drug: Atazanavir 300mg/ Ritonavir 100 mg once daily

INTERVENTIONS:
Drug: Atazanavir 300mg/ Ritonavir 100 mg once daily — There is no intervention in this study - participants will all be receiving atazanavir (usually boosted with ritonavir) as part of their routine clinical care
  Groups: Adolescents 12-17; BMI < 18.5; BMI >30; Pregnant women
Drug: Atazanavir 250 mg / ritonavir 80 mg — There is no intervention in this study - participants will all be receiving atazanavir (usually boosted with ritonavir) as part of their routine clinical care. This dose of 250/ 80 is for participants weighing between 15 and 25 Kg
  Groups: Children 6-11; Children <5 years

SUMMARY:
The lack of data relating to the DDI between ATV and RIF is a major limitation to the use of ATV in patients who require treatment for TB. The VirTUAL Workpackage 2 will explore the necessary dose escalation required to overcome this interaction in non-pregnant HIV-infected adults who are virologically suppressed on bPI-based ART, and who are administered RIF as a study drug, not as part of a full TB treatment regimen. As the specific objective of WP2 is to define the dose of ATV, participants taking an alternative bPI will be transitioned to ATV for the duration of that study. However, to extrapolate the results of this study to special populations such as pregnant and postpartum women, children and adolescents and those with other 'special' characteristics such as obesity (BMI >30 Kg/m2) or malnutrition (BMI <18.5 Kg/m2) we propose to undertake sparse sampling for pharmacokinetic analysis from individuals who require ATV-based ART for their clinical care.

Sparse PK data will be obtained opportunistically from participants in the 'special populations' defined above who are receiving ATV as part of their routine clinical care. Subjects will be identified from clinics including the Joint Clinical Research Center (JCRC) and Infectious Diseases Institute (IDI), Kampala, and from sites including Groote Schuur Hospital and Gugulethu Community Health Centre, Cape Town. The ATV/r data from "special populations" will enable validation and refinement of both the PBPK model (WP1) and the pop-PK models (WP4) of the VirTUAL consortium.

DETAILED DESCRIPTION:
Overview of VirTUAL Consortium Through the VirTUAL Consortium, the investigators aim to define the optimal use of second-line ART regimens in vulnerable populations with TB co-infection. The primary objective is to 'to determine the optimal dose of boosted atazanavir (ATV/r) when used in combination with RIF-based TB treatment in children, adolescents and pregnant or breastfeeding women.'

The results from this protocol (VirTUAL WP5) will be considered in the context of the full research programme. This can be summarised as follows:

Physiologically-based pharmacokinetic (PBPK) modelling will be developed to understand bPI and RIF Drug-Drug Interactions (DDIs), identifying potential dosing strategies to overcome these in adults and special populations (WP1). This data will inform clinical pharmacokinetic studies exploring the necessary dose escalation of ATV/r, including in the context of high-dose RIF, performed in Kampala (WP2). Intracellular pharmacokinetics will further characterise the DDI (WP3). PBPK and population pharmacokinetics (pop-PK) modelling will be integrated enabling extrapolation to special populations (WP4), and sparse data collection from such populations receiving different combinations of second-line ART and/or TB treatment in Kampala and Cape Town will validate and refine these models (WP5). Capacity building focussing on equipping African scientists with the tools to efficiently define drug dosing in complex populations (WP6), communication and stakeholder engagement (WP7) will increase the application of this methodology to other priority research into pharmacokinetics in special populations.

This protocol describes the sparse pharmacokinetic sampling component which forms Workpackage 5 (WP5) of this research programme. The dose-escalation study (WP2) is an interventional trial which will be conducted in 28 healthy, virologically suppressed volunteers who are on ATV-based second-line ART, are aged over 18, have a normal BMI and are not pregnant or breastfeeding, and which will take place at JCRC, Kampala, Uganda. This study is anticipated to commence in mid-2019, and will explore in detail the changes in pharmacokinetics of ATV/r in both plasma and within cells which take place when rifampicin is co-administered, and will evaluate the necessary dose adjustment which is required to concurrently administer ATV/r with rifampicin-based TB treatment. WP2 will generate intensive data on these 28 well characterized individuals who do not have 'special' characteristics. However, there is a paucity of data on ATV/r disposition in patients who are typically excluded from clinical trials, and therefore the observational data from WP5 will be collected from individuals who fall into the listed categories of special populations and who are being treated with ATV/r for their own health. Data from either WP2 or WP5 alone will be amenable to pharmacometric analysis and bring value, but the combined modelling approach using both sets of data in a combined model will allow the most comprehensive evaluation of ATV/r disposition in the wider population, and will enable projections of dosing recommendations for the special populations who require concurrent treatment for TB whilst receiving ATV/r-based ART.

Individuals will be identified at routine clinic appointments. They (or their guardians) will be asked to keep a detailed record of dosing times for three to five days prior to their study appointment at which sampling will be performed. If they take their medication in the morning, they will be asked to bring the medication to clinic for observation of dosing.

Repeat sampling at subsequent appointments will enable assessment of both between and within-individual variability, for example during periods of rapid childhood growth or during pregnancy and transition back to non-pregnant physiological state.

It is aimed to obtain 20 sparse PK profiles in each of the following groups (pregnant, child <5, child 6-11, adolescent 12-18, obese (BMI >30 Kg/m2), malnourished (BMI <18.5 Kg/m2)), with each individual contributing 4 samples per PK visit, and possibly followed up longitudinally during the study (each individual may attend for a maximum of three study visits). Therefore there will be between 7 (6 participants being sampled on 3 occasions and a final participant sampled on 2 occasions) and 20 (if each participant was only sampled on a single occasion) individual participants per group to generate the 20 sampling 'occasions', with a total number of participants across the six groups included in the study of between 42 and 120.

This will provide an essential clinical dataset to inform the pop-PK modelling approach and validate the PBPK simulations, describing exposure and pharmacokinetic variability in the populations of interest. The data from this work package will be pooled with the data from the study in volunteers and jointly analysed using PK modelling. Differences in the PK parameters for each of the groups will be investigated.

There exist no peer-reviewed published data regarding the transfer of ATV/r into breast milk. Therefore, among women who are enrolled during pregnancy and followed into the postpartum phase, paired breast milk samples will be obtained at the same time as plasma samples.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the participant (or a legal representative) has been informed of all pertinent aspects of the study.
2. In a child aged ≥7 years (South Africa) or aged ≥8 years (Uganda), evidence of assent to participate
3. Participants who are willing and able to comply with scheduled visits, laboratory tests, and other study procedures.
4. HIV-infected, receiving ATV-based ART treatment OR HIV-infected receiving second-line ART with concurrent rifamycin-based TB treatment
5. Participant is within one of the target populations:

   1. Pregnant (>20 weeks)
   2. Body mass index >30 or <18.5 Kg/m2
   3. Child or adolescent aged <18 years

Exclusion Criteria:

1. Medical, psychiatric or obstetric condition that might affect participation in the stuy based on investigator judgement
2. Dissent from a minor
3. For pregnant women in Uganda, where the husband is reasonably involved, paternal objection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — One of the groups of special interest is pregnant women, who will all be female
Study Population: Individuals will be identified at routine clinic appointments. They (or their guardians) will be asked to keep a detailed record of dosing times for three to five days prior to their study appointment at which sampling will be performed. If they take their medication in the morning, they will be asked to bring the medication to clinic for observation of dosing.
  Repeat sampling at subsequent appointments will enable assessment of both between and within-individual variability, for example during periods of rapid childhood growth or during pregnancy and transition back to non-pregnant physiological state.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Atazanavir Cmax | 3 years
  To describe the maximum concentration of atazanavir reached after dosing in the different groups
Atazanavir AUC0-24 | 3 years
  To describe the area under the concentration-time curve from 0 to 24 hours after dosing in the different groups
Atazanavir Ctau | 3 years
  To describe the trough concentration of atazanavir after dosing in the different study groups

SECONDARY OUTCOMES:
Comparison of geometric mean of atazanavir Cmax with healthy adult population | 3 years
  To compare atazanavir Cmax with typical healthy individuals treated with atazanavir who enter a dose escalation study of ATV/r + RIF as WP2 of the VirTUAL programme
Comparison of geometric mean of atazanavir AUC0-24 with healthy adult population | 3 years
  To compare atazanavir AUC0-24 with that of typical healthy adults treated with atazanavir-based ART who enter a dose escalation study of ATV/r + RIF as WP2 of the VirTUAL programme
Comparison of geometric mean of atazanavir Ctau with healthy adult population | 3 years
  To compare atazanavir Ctau with that of typical healthy adults treated with atazanavir-based ART who enter a dose escalation study of ATV/r + RIF as WP2 of the VirTUAL programme

OTHER OUTCOMES:
Modelling of atazanavir pharmacokinetics | 4 years
  To use nonlinear mixed-effects modelling to describe sources of variability on the pharmacokinetics of ATV
Exploratory objective: Cmax of second-line ART with TB treatment | 3 years
  To describe the maximum concentrations of second-line antiretroviral drugs and rifamycin-containing TB therapy in HIV-infected pregnant and postpartum women, children and adolescents and individuals with extremes of BMI
Exploratory objective: AUC of second-line ART with TB treatment | 3 years
  To describe the area under the concentration-time curve of second-line antiretroviral drugs and rifamycin-containing TB therapy in HIV-infected pregnant and postpartum women, children and adolescents and individuals with extremes of BMI
Exploratory objective: Ctau of second-line ART with TB treatment | 3 years
  To describe the minimum concentration of second-line antiretroviral drugs and rifamycin-containing TB therapy in HIV-infected pregnant and postpartum women, children and adolescents and individuals with extremes of BMI

CONTACTS AND LOCATIONS:
Locations (4):
- South Africa (2):
  - Desmond Tutu HIV Foundation, Cape Town, Western Cape
  - University of Cape Town, Cape Town, Western Cape
- Uganda (2):
  - Infectious Diseases Institute, Kampala
  - Joint Clinical Research Centre, Kampala

IPD SHARING:
Plan to Share IPD: No